CLINICAL TRIAL: NCT02267603
Title: A Phase II Study of MK-3475 in Patients With Advanced Merkel Cell Carcinoma (MCC)
Brief Title: Pembrolizumab in Treating Patients With Advanced Merkel Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-00848; NCI-2014-00848 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MK-3475; CITN-09; CITN-09 (Other: Cancer Immunotherapy Trials Network); CITN-09 (Other: CTEP); K24CA139052 (NIH); P30CA015704 (NIH); U01CA154967 (NIH)
Record Dates: First submitted 2014-10-14; First posted 2014-10-17 (Estimated); Results first posted 2019-03-01 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Recurrent Merkel Cell Carcinoma; Stage III Merkel Cell Carcinoma AJCC v7; Stage IIIA Merkel Cell Carcinoma AJCC v7; Stage IIIB Merkel Cell Carcinoma AJCC v7; Stage IV Merkel Cell Carcinoma AJCC v7
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 24 months in the absence of disease progression* or unacceptable toxicity.
  * NOTE: Patients with confirmed disease progression may continue to receive treatment if they are otherwise clinically stable until there is an increase in tumor burden of 25% or more following initial confirmation of progression. Under exceptional circumstances, and with protocol P.I. and CITN P.I. approval, patients may receive treatment beyond 2 years.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Ancillary studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab works in treating patients with Merkel cell cancer that cannot be removed by surgery or controlled with treatment, or has spread to other parts of the body. Pembrolizumab may stimulate the immune system to identify and destroy cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the clinical efficacy of MK-3475 (pembrolizumab) as the first systemic intervention for patients with advanced Merkel cell carcinoma (MCC).

SECONDARY OBJECTIVES:

I. To determine the clinical activity of MK-3475 as the first systemic intervention for patients with advanced MCC.

TERTIARY OBJECTIVES:

I. To determine the immune correlates of the clinical activity of MK-3475.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 21 days for up to 24 months in the absence of disease progression* or unacceptable toxicity.

* NOTE: Patients with confirmed disease progression may continue to receive treatment if they are otherwise clinically stable until there is an increase in tumor burden of 25% or more following initial confirmation of progression. Under exceptional circumstances, and with protocol principal investigator (P.I.) and Cancer Immunotherapy Trials Network (CITN) P.I. approval, patients may receive treatment beyond 2 years.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for 1 year, every 6 months for 2 years, annually until the patient has completed 3 years of follow up for disease assessment, and then every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have biopsy-proven metastatic MCC or locoregional MCC that has recurred following standard locoregional therapy with surgery and/or radiation therapy
* Patients must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 assessed by computed tomography (CT) scan, or for skin lesions not measurable by CT scan, measurements may be performed with caliper or flexible ruler

  * Note: stage IV no evidence of disease (NED) is excluded by this criterion
* Have a performance status of =< 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Life expectancy of greater than 6 months
* Leukocytes >= 2,000/mcL (labs should be performed within 14 days of treatment initiation)
* Absolute neutrophil count >= 1,500/mcL (labs should be performed within 14 days of treatment initiation)
* Platelets >= 100,000/mcL (labs should be performed within 14 days of treatment initiation)
* Hemoglobin >= 9 g/dL OR >= 5.6 mmol/L (labs should be performed within 14 days of treatment initiation)
* Serum total bilirubin =< 1.5 x upper limit of normal (ULN) OR direct bilirubin =< ULN for patients with total bilirubin levels > 1.5 x ULN (labs should be performed within 14 days of treatment initiation)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN OR =< 5 x ULN for patients with liver metastases (labs should be performed within 14 days of treatment initiation)
* Serum creatinine =< 2.5 x ULN OR measured or calculated* creatinine clearance (CrCl) (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 30 mL/min for subject with creatinine levels > 2.5 x institutional ULN

  * Creatinine clearance should be calculated per institutional standard (labs should be performed within 14 days of treatment initiation)
* Thyroid stimulating hormone (TSH) within institutional limits (i.e.: normal); if TSH is greater or less than institutional limits patients may participate if their T4 is within normal limits (WNL); patients may be on a stable dose of replacement thyroid medication; dose adjustments are allowed if needed (labs should be performed within 14 days of treatment initiation)
* Patients must provide tissue from an archival tumor sample or newly obtained core, punch or excisional biopsy of a tumor lesion if deemed relatively safe and technically feasible

  * Note: newly obtained biopsy is preferable
* Female patients of childbearing potential must have a negative urine or serum pregnancy within 72 hours before receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required

  * Note: women of child-bearing potential must agree to use 2 methods of birth control, or be surgically sterile, or abstain from heterosexual activity beginning with the screening visit and for the duration of study participation, through 120 days beyond last dose of MK-3475 administration; patients of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Men treated or enrolled on this protocol must agree to use 2 adequate methods of contraception starting with the screening visit, for the duration of study participation, and through 120 days after the last dose of MK-3475 administration
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Patient has had prior systemic therapy for MCC

  * Note: prior systemic cytotoxic chemotherapy will be allowed if it was administered in the adjuvant setting (no clinically detectable MCC at the time) and treatment concluded more than 6 months prior to beginning study treatment
* Patient is currently participating in or has participated in a study of an investigational systemic agent to treat MCC; or is using an investigational device within 4 weeks of the first dose of treatment

  * NOTE: if patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
  * Toxicity from surgery or associated interventions that has not recovered to =< grade 1 is allowed if it meets the inclusion requirements for laboratory parameters
* Patients with locoregional disease that have not received appropriate standard locoregional therapy with surgery and/or radiation therapy
* Patient has had radiation therapy within 2 weeks of beginning study treatment
* Toxicity from prior radiation therapy has NOT resolved to grade 1 or less
* Patient has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior the first dose of trial treatment
* Patient has had a prior monoclonal antibody for treatment of MCC
* Patient has had a prior monoclonal antibody for a non-cancer therapy indication within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events (AEs) due to agents administered more than 4 weeks earlier
* Patient has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Patient has known active central nervous system (CNS) metastases and/or carcinomatous meningitis

  * Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment
* Patient has a history of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-3475
* Patient has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents; patients with vitiligo or resolved childhood asthma/atopy would be an exception to this rule; patients that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study; the use of physiologic doses of corticosteroids may be approved after consultation with the protocol principal investigator (PI) and Cancer Immunotherapy Trials Network (CITN); patients with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study
* Patient has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator
* Patient has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Patient has uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, interstitial lung disease, non-infectious pneumonitis, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patient is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment

  * NOTE: pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with MK-3475
  * Men and nonpregnant, non-breast-feeding women may be enrolled if they are willing to use 2 methods of birth control or are considered highly unlikely to conceive; highly unlikely to conceive is defined as (1) surgically sterilized, or (2) postmenopausal (a woman who is >= 45 years of age and has not had menses for greater than 1 year will be considered postmenopausal), or (3) not heterosexually active for the duration of the study; the 2 birth control methods can be barrier method or a barrier method plus a hormonal method to prevent pregnancy; subjects should start using birth control from the screening visit throughout the study period up to 120 days after the last dose of study therapy
  * The following are considered adequate barrier methods of contraception: diaphragm, condom (by the partner), copper intrauterine device, sponge, or spermicide; appropriate hormonal contraceptives will include any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent (including oral, subcutaneous, intrauterine, or intramuscular agents)
  * Patients should be informed that taking the study medication may involve unknown risks to the fetus (unborn baby) if pregnancy were to occur during the study; in order to participate in the study, they must adhere to the contraception requirement (described above) for the duration of the study and during the follow-up period described above; if there is any question that a subject will not reliably comply with the requirements for contraception, that subject should not be entered into the study
  * Pregnancy: if a patient inadvertently becomes pregnant while on treatment with MK-3475, the patient will immediately be removed from the study; the site will contact the patient at least monthly and document the patient's status until the pregnancy has been completed or terminated; the outcome of the pregnancy will be reported without delay and within 24 hours if the outcome is a serious adverse experience (e.g., death, abortion, congenital anomaly, or other disabling or life-threatening complication to the mother or newborn); the study investigator will make every effort to obtain permission to follow the outcome of the pregnancy and report the condition of the fetus or newborn; if a male patient impregnates his female partner the study personnel at the site must be informed immediately and the pregnancy reported and followed
  * Subjects who are breast-feeding are not eligible for enrollment
* Patient is human immunodeficiency virus (HIV) positive

Note: patients who are human immunodeficiency virus (HIV) positive may participate IF they meet the following eligibility requirements:

* They must be stable on their anti-retroviral regimen, and they must be healthy from an HIV perspective
* They must have a cluster of differentiation (CD)4 count of greater than 250 cells/mcL
* They must not be receiving prophylactic therapy for an opportunistic infection

  * Patient has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Note: a positive hepatitis B serology indicative of previous immunization (i.e., hepatitis B surface antibody [HBsAb]-positive and hepatitis B core antibody [HBcAb]-negative) or a fully resolved acute hepatitis B infection is not an exclusion criterion

  * Has active non-infectious pneumonitis >= grade 2; or history of grade 3 non-infectious pneumonitis within the past 12 months; or any history of grade 4 non-infectious pneumonitis
  * History of other pulmonary disease such as emphysema or chronic obstructive pulmonary disease (COPD), (forced expiratory volume in 1 second [FEV1] < 60% of predicted for height and age); pulmonary function tests (PFTs) are required in patients with prolonged smoking history or symptoms of respiratory dysfunction
  * Cardiovascular disease that meets one of the following: congestive heart failure (New York Heart Association class III or IV), active angina pectoris, or recent myocardial infarction (within the last 6 months)
  * Prior organ allograft or allogeneic transplantation, if the transplanted tissue is still in place
  * Patient has had live vaccines within 30 days before the first dose of trial treatment and while participating in the trial; examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, seasonal flu, H1N1 flu, rabies, bacille de Calmette et Guérin (BCG), and typhoid vaccine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-11-25 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2021-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Nghiem, Principal Investigator — Cancer Immunotherapy Trials Network
Locations (13):
- United States (13):
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Mount Sinai Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Seattle Cancer Care Alliance, Seattle, Washington

REFERENCES:
- [Derived] Nghiem P, Bhatia S, Lipson EJ, Sharfman WH, Kudchadkar RR, Brohl AS, Friedlander PA, Daud A, Kluger HM, Reddy SA, Boulmay BC, Riker A, Burgess MA, Hanks BA, Olencki T, Kendra K, Church C, Akaike T, Ramchurren N, Shinohara MM, Salim B, Taube JM, Jensen E, Kalabis M, Fling SP, Homet Moreno B, Sharon E, Cheever MA, Topalian SL. Three-year survival, correlates and salvage therapies in patients receiving first-line pembrolizumab for advanced Merkel cell carcinoma. J Immunother Cancer. 2021 Apr;9(4):e002478. doi: 10.1136/jitc-2021-002478. PMID 33879601
- [Derived] Nghiem P, Bhatia S, Lipson EJ, Sharfman WH, Kudchadkar RR, Brohl AS, Friedlander PA, Daud A, Kluger HM, Reddy SA, Boulmay BC, Riker AI, Burgess MA, Hanks BA, Olencki T, Margolin K, Lundgren LM, Soni A, Ramchurren N, Church C, Park SY, Shinohara MM, Salim B, Taube JM, Bird SR, Ibrahim N, Fling SP, Homet Moreno B, Sharon E, Cheever MA, Topalian SL. Durable Tumor Regression and Overall Survival in Patients With Advanced Merkel Cell Carcinoma Receiving Pembrolizumab as First-Line Therapy. J Clin Oncol. 2019 Mar 20;37(9):693-702. doi: 10.1200/JCO.18.01896. Epub 2019 Feb 6. PMID 30726175
- [Derived] Nghiem PT, Bhatia S, Lipson EJ, Kudchadkar RR, Miller NJ, Annamalai L, Berry S, Chartash EK, Daud A, Fling SP, Friedlander PA, Kluger HM, Kohrt HE, Lundgren L, Margolin K, Mitchell A, Olencki T, Pardoll DM, Reddy SA, Shantha EM, Sharfman WH, Sharon E, Shemanski LR, Shinohara MM, Sunshine JC, Taube JM, Thompson JA, Townson SM, Yearley JH, Topalian SL, Cheever MA. PD-1 Blockade with Pembrolizumab in Advanced Merkel-Cell Carcinoma. N Engl J Med. 2016 Jun 30;374(26):2542-52. doi: 10.1056/NEJMoa1603702. Epub 2016 Apr 19. PMID 27093365

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was expanded from 24 patients to 50 patients at the request of the pharmaceutical collaborator.
Groups:
- Treatment (Pembrolizumab): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 24 months in the absence of disease progression* or unacceptable toxicity.
  * NOTE: Patients with confirmed disease progression may continue to receive treatment if they are otherwise clinically stable until there is an increase in tumor burden of 25% or more following initial confirmation of progression. Under exceptional circumstances, and with protocol P.I. and CITN P.I. approval, patients may receive treatment beyond 2 years.
  Laboratory Biomarker Analysis: Ancillary studies
  Pembrolizumab: Given IV
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab)
Started | 50
Completed | 6
Not Completed | 44

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 45
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Defined as the Proportion of Patients Who Have Achieved Complete Response (CR) or Partial Response (PR) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: ORR will be estimated as the number of responders as a percent of the number of eligible participants who received at least one dose of treatment. If a substantial amount of data is missing, analyses will be performed using parametric generalized linear models fit by maximum likelihood. A generalized linear model for the ORR will use a binomial error distribution. The model will include as covariates all available baseline predictors of the missing outcomes. Responses to continued pembrolizumab will be chronicled and reported.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 50
Participants
  Number participants with partial response (PR) | 16
  Number participants with complete response (CR) | 12
  Combined total participants with either PR or CR | 28
Statistical Analysis 1: Comparison: Treatment (Pembrolizumab); The protocol was designed w/ a standard Simon 2 stage design. Null hypothesis that true response rate is 5% was tested against a 1-sided alternative. In stage 1, 9 patients were accrued. If no responses in these 9 patients, study was to stop. Otherwise,15 more patients were to be accrued for a total of 24 patients. Study was amended to increase number of patients to 50, following discussion w/ pharmaceutical collaborator and FDA; Test type: Other — The null hypothesis will be rejected if 3 or more responses are observed in 24 patients. This design yields a type I error rate of 0.10 and power of 0.90 when the true response rate is 25%. Progression-free survival (PFS) at 16 months will be estimated by Kaplan-Meier method. Unless otherwise stated, all statistical tests will be conducted at the α=0.05 (1-sided) level; ORR will be estimated as the # of responders as a % of the # of eligible participants who received at least 1 dose of treatment. If a substantial amount of primary endpoint data are missing (at least 1 value missing from more than 20% of participants), using nonparametric estimation to estimate the ORR requires the missing completely at random assumption may give misleading results. In this case, analyses of the primary endpoint will be performed using parametric generalized linear models fit by maximum likelihood. These methods provide unbiased estimation and inferences under the parametric modeling assumptions and the assumption that the missing data are missing at random (MAR). MAR assumes that the probability of an observation being missing may depend upon the observed responses and upon observed covariates. A generalized linear model for the ORR will use a binomial error distribution. The model will include as covariates all available baseline predictors of the missing outcomes

2. Secondary Outcome: Progression-free Survival (PFS) Using RECIST 1.1
Description: Survival curves for PFS will be estimated using the Kaplan-Meier method. Assessed percentage of participants with progression free survival up to 16 months.
Time Frame: Time from start of treatment to time of progression or death, whichever occurs first, assessed up to 16 months
Measure: Number; unit: % of participants
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 50
% of participants | 49.9

3. Secondary Outcome: Duration of Response (DOR)
Description: Survival curves for DOR will be estimated using the Kaplan-Meier method.
Time Frame: Time interval between the date of first response (CR/PR) and the date of progression, assessed up to 3 years
Population: Thirty participants with durable response were assessed by RECIST 1.1.
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 30
months | NA [4.0 to 77.4] — Median was not reached due to insufficient number of events, i.e., (too few participants had reached progression at data cutoff.)

4. Secondary Outcome: Overall Survival (OS)
Description: Survival curves for OS will be estimated using the Kaplan-Meier method.
Time Frame: Time interval between the start of treatment to death due to any cause, assessed up to 60 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 50
months | 47.2 [26 to 68.4]

5. Secondary Outcome: Incidence of Adverse Events (AEs) Graded Using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Description: Safety will be assessed by quantifying the toxicities and grades experienced by subjects including serious AEs (SAEs) and events of clinical interest. Safety and tolerability will be assessed by clinical review of all relevant parameters including AEs, laboratory tests, vital signs, and electrocardiogram measurements. Assessed number of participants who experienced grade 3 to 5 adverse events.
Time Frame: Up to 90 days post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 50
Participants
  Grade 3-5 Adverse Events | 29
  Grade 3-5 Drug Related Adverse Events | 15

6. Other Pre Specified Outcome: Immune Correlates of the Clinical Activity of Pembrolizumab
Description: This will include immunohistochemical and gene expression analysis focusing on delineating the immune components and immunologic milieu within the tumor before therapy.
Time Frame: Baseline
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Merkel Polyomavirus (MCPyV)-Specific Immune Response, Assessed With Enzyme-linked Immunosorbent Spot and Serology Assays
Description: Responses will be assessed at baseline, after initiating therapy, and correlated with clinical responses over time. Among patients with corresponding MHC-peptide tetramers, pre- and post-treatment samples of circulating MCPyV-specific CD8 T cells will be isolated and subjected to deep immunophenotyping by messenger ribonucleic acid (mRNA) expression analysis.
Time Frame: After 2 years of treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Serious Adverse Events and other (not including serious) adverse events were assessed for up to 36 months. All cause mortality was assessed for up to 60 months.
Arm/Group | Treatment (Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 16/50
Serious Adverse Events (participants affected / at risk) | 22/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Pembrolizumab) (N=50)
Anemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Myocarditis (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Chills (General disorders) | 1
Disease progression (General disorders) | 8
Fatigue (General disorders) | 2
Malaise (General disorders) | 1
Pyrexia (General disorders) | 2
Lung infection (Infections and infestations) | 1
Mastitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sialoadenitis (Infections and infestations) | 1
Streptococcal bacteraemia (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Delirium (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Embolism (Vascular disorders) | 3
Haematoma (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Pembrolizumab) (N=50)
Anaemia (Blood and lymphatic system disorders) | 16
Leukocytosis (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 2
Lymph node pain (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 1
Monocytosis (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Bundle branch block left (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Deafness (Ear and labyrinth disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 2
Paraesthesia ear (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 1
Autoimmune hypothyroidism (Endocrine disorders) | 2
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 3
Thyroiditis (Endocrine disorders) | 1
Asthenopia (Eye disorders) | 1
Diplopia (Eye disorders) | 1
Eyelid ptosis (Eye disorders) | 1
Ophthalmoplegia (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Visual impairment (Eye disorders) | 2
Vitreous floaters (Eye disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 2
Aphthous ulcer (Gastrointestinal disorders) | 1
Breath odour (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 14
Diarrhoea (Gastrointestinal disorders) | 11
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Faeces discoloured (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4
Haemorrhoids (Gastrointestinal disorders) | 1
Intra-abdominal haematoma (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 10
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 2
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Chills (General disorders) | 4
Cyst (General disorders) | 1
Face oedema (General disorders) | 1
Fatigue (General disorders) | 28
Feeling cold (General disorders) | 1
Feeling hot (General disorders) | 2
Gait disturbance (General disorders) | 1
Malaise (General disorders) | 1
Nodule (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 4
Pain (General disorders) | 1
Peripheral swelling (General disorders) | 4
Pyrexia (General disorders) | 7
Swelling (General disorders) | 2
Temperature intolerance (General disorders) | 2
Autoimmune hepatitis (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Abdominal hernia infection (Infections and infestations) | 1
Abscess limb (Infections and infestations) | 1
Breast cellulitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 3
Conjunctivitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Eye infection (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 1
Genital herpes (Infections and infestations) | 1
Herpes virus infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 4
Lung infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 3
Oral candidiasis (Infections and infestations) | 3
Oral herpes (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 3
Skin infection (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Streptococcal infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 14
Urinary tract infection (Infections and infestations) | 6
Vaginal infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 3
Excoriation (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 11
Amylase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 8
Blood alkaline phosphatase decreased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 7
Blood bilirubin increased (Investigations) | 4
Blood creatine phosphokinase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 6
Blood glucose increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Blood magnesium increased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Blood testosterone decreased (Investigations) | 1
Blood thyroid stimulating hormone increased (Investigations) | 1
Blood urea increased (Investigations) | 1
Blood urine present (Investigations) | 1
Lipase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 7
Neutrophil count decreased (Investigations) | 1
Neutrophil count increased (Investigations) | 1
Platelet count decreased (Investigations) | 2
Sputum normal (Investigations) | 1
Thyroxine free increased (Investigations) | 2
Weight decreased (Investigations) | 5
White blood cell count decreased (Investigations) | 5
Decreased appetite (Metabolism and nutrition disorders) | 11
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2
Hyperchloraemia (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 11
Hyperkalaemia (Metabolism and nutrition disorders) | 4
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 7
Hypochloraemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 10
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Hypoproteinaemia (Metabolism and nutrition disorders) | 2
Hypovitaminosis (Metabolism and nutrition disorders) | 1
Increased appetite (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Neck mass (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Burning sensation (Nervous system disorders) | 2
Cerebral ischaemia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 8
Dysgeusia (Nervous system disorders) | 4
Encephalopathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 10
Hyperaesthesia (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 3
Lethargy (Nervous system disorders) | 2
Memory impairment (Nervous system disorders) | 1
Nystagmus (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 3
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 3
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Disorientation (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Irritability (Psychiatric disorders) | 2
Mental status changes (Psychiatric disorders) | 2
Mood altered (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 4
Acute kidney injury (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 2
Glycosuria (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 3
Nephritis (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Breast pain (Reproductive system and breast disorders) | 3
Breast swelling (Reproductive system and breast disorders) | 2
Oedema genital (Reproductive system and breast disorders) | 1
Pruritus genital (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1
Hypotrichosis (Skin and subcutaneous tissue disorders) | 1
Itching scar (Skin and subcutaneous tissue disorders) | 1
Lichen planus (Skin and subcutaneous tissue disorders) | 1
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 2
Night sweats (Skin and subcutaneous tissue disorders) | 2
Papule (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 11
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 11
Rash erythematous (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7
Rash pruritic (Skin and subcutaneous tissue disorders) | 2
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Cancer surgery (Surgical and medical procedures) | 1
Cataract operation (Surgical and medical procedures) | 1
Deep vein thrombosis (Vascular disorders) | 1
Embolism (Vascular disorders) | 1
Haematoma (Vascular disorders) | 2
Hot flush (Vascular disorders) | 5
Hypertension (Vascular disorders) | 6
Hypotension (Vascular disorders) | 4
Lymphoedema (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/03/NCT02267603/Prot_SAP_000.pdf